CLINICAL TRIAL: NCT06897943
Title: Epidemiology of Gonococcal Arthritis
Brief Title: Epidemiology of Gonococcal Arthritis (EpGAr)
Acronym: EpGAr
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0339 - EpGAr
Record Dates: First submitted 2025-03-10; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Gonococcal (GC) Infection; Arthritis, Infectious
Keywords: gonococcal arthritis
MeSH Terms: conditions — Gonorrhea; Infections; Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gonococcal arthritis: Patients with a positive joint sample for Neisseria gonorrhoeae between 06/01/2014 and 06/30/2024 in Brittany, France.

SUMMARY:
The aim of this retrospective observational study was to describe the epidemiology of Neisseria gonorrhoeae septic arthritis over the last 10 years at Brest and Rennes university hospitals. The main question is whether there are any risk factors based on the epidemiological and clinical data on these cases. The second objective is to characterize the gonococcal strains isolated in order to determine whether there is a common clone, a virulence factor or specific resistance genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Neisseria gonorrhoeae-positive joint sample (from an enrichment vial or a native sample) between 2014 and 2024.

Exclusion Criteria:

* Patients with Neisseria gonorrhoeae-negative joint sample (from enrichment vial or native sample).
* Patients who have expressed opposition to inclusion in the study.
* Patients under legal protection (guardianship, curatorship, etc.).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a Neisseria gonorrhoeae-positive joint sample (from an enrichment vial or a native sample) between 06/01/2014 and 06/30/2024.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Age | 10 years
  years
Date of sampling | 10 years
  DD/MM/YYYY
Type of sample | 10 years
  joint fluid or joint fluid on blood culture bottle
Rate of white blood cells | 10 years
  quantification of white blood cells /mm3
Sexually transmitted infection | 10 years
  associated or not, if associated, name of STI and localization
Men who have sex with men | 10 years
  yes or no
HIV pre-exposure prophylaxis (PreP) | 10 years
  yes or no
Comorbidities | 10 years
  any history mentioned in the medical file, such as fracture, illness, treatment, chronic alcoholism, cancer, diabetes, etc.
Imaging | 10 years
  medical conclusion of the ultrasound or radiology performed
Blood cultures (peripheral blood) | 10 years
  positive or negative
Time to diagnosis | 10 years
  in days (between onset of symptoms and antibiotics)
Treatments implemented | 10 years
  name of the probabilistic treatment (antibiotic) and after identification or antibiogram
Antibiotic sensitivity profile | 10 years
  Susceptibility or resistance according to SIR methodology and, if achieved: minimum inhibitory concentrations of antibiotics tested on the strain in mg/L
Surgery | 10 years
  yes or not
Evolution | 10 years
  recovery or relapse
Rate of neutrophils | 10 years
  proportion of neutrophils in %.
Rate of CRP (C-reactive protein) | 10 years
  in mg/L

SECONDARY OUTCOMES:
Molecular typing: clone | 10 years
  performed on strains sent to the Centre National de Référence des IST - APHP
Molecular typing: virulence factors | 10 years
  performed on strains sent to the Centre National de Référence des IST - APHP
Molecular typing: resistance genes | 10 years
  performed on strains sent to the Centre National de Référence des IST - APHP

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève HERY-ARNAUD, Principal Investigator — CHU de Brest
Locations (2):
- France (2):
  - Rennes University Hospital, Rennes, Brittany Region
  - CHU de BREST, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement